CLINICAL TRIAL: NCT04749966
Title: Understanding Wellbeing Among Emergency Service Staff by Mapping Physiological Indicators and Subjective Mediators of Stress: An Observational Feasibility Study
Brief Title: Blue Light Emergency Services Wellbeing Feasibility Study
Status: Completed | Type: Observational
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Other Study IDs: 19_20_029; IRAS 278059 (Other: UK Health Research Authority)
Record Dates: First submitted 2021-01-29; First posted 2021-02-11 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-10

CONDITIONS: Wellbeing
Keywords: Emergency services; wellbeing; stress; physiological responses; subjective mediators

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency services staff: Emergency Services staff recruited from the Ambulance, Police, and Fire and Rescue Services.
  Interventions: Other: This is an observational study, there are no interventions

INTERVENTIONS:
Other: This is an observational study, there are no interventions — This is an observational study, there are no interventions

SUMMARY:
Emergency Service teams operate in some of the most challenging workplaces and experience higher rates of mental ill health than the general population. Effective interventions are required to enhance wellbeing, but as a first step it is crucial to understand the context through which to develop these initiatives. This preliminary study will test the feasibility of implementing a larger study to map the relationship between physical responses associated with levels of stress (heart rate variability) and personal, social and organisational factors that mediate these responses. In doing so, it is hoped to provide an insight into factors that shape emergency staff members' response to stress to help develop and personalise wellbeing initiatives.

DETAILED DESCRIPTION:
The study team is proposing a large study in the Essex Emergency Services to map the relationship between physiological indicators of stress and subjective mediators and, in doing, provide insight into factors that shape a staff members' response to stress, which could help to develop and personalise wellbeing initiatives.

However, before undertaking a large study it is proposed to establish operational feasibility. This feasibility study will enrol ten shift-working staff from each of three emergency services (Essex Police, Essex County Fire and Rescue Service and East of England Ambulance Service Trust). Over a 3-day period, we will evaluate participants' physiological response to stressors by measuring HRV (using Firstbeat Bodyguard 2 beat-to-beat heart rate monitor). During the same period, participants will keep a personal online journal of events during the day. As part of the lifestyle assessment, data from the heart rate monitor and journal will be analysed and participants will receive a Summary Report including information on their body's reaction to stress and how this may be managed. Following the lifestyle assessment, the research team will facilitate semi-structured interviews; they will use participants' lifestyle assessment Summary Reports to inform appropriate questions. The team will discuss subjective experiences with participants as well as their overall experience with the data collection process.

The objectives of the feasibility study are to:

1. Evaluate feasibility of undertaking a larger definitive study in terms of:

   * Willingness and eligibility of emergency services' staff to take part in the study
   * Recruitment timeframe
   * Participant adherence to lifestyle assessment protocols (including wearing a heart rate monitor and completing an online journal over a 3-day period)
   * Proportion of participants in whom an interview is arranged and completed
   * Feasibility of other operational aspects not included above.
2. Undertake an initial evaluation of physiological indicators and subjective mediators of stress and identify any i) associations between them and ii) patterns that emerge between individual participants.

ELIGIBILITY:
Inclusion Criteria:

* are aged 18 or older
* full-time employees
* work shift patterns and will be on-duty during the study period
* are able to take part in and contribute to the study (see exclusion criteria below).

Exclusion Criteria:

* off-duty or on leave during the study period
* part-time (or on-call) employees
* not working shift patterns
* currently taking part in research that may impact on results, design or scientific value of this study (or other studies)
* not able to read or understand the English Language as it will not be possible to provide translation services for the study

In addition, the results from the heart rate monitor may be unreliable with certain medical conditions and, as such, staff will not be able to take part if they have had a heart transplant or if they have a pacemaker, heart disease, atrial fibrillation, atrial flutter or uncontrolled thyroid disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A purposive, non-probability sample will be selected and recruited comprising ten operational shift working staff from each of three emergency services (Essex Police, Essex County Fire and Rescue Service and East of England Ambulance Trust).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of study recruitment - the number of staff volunteering to take part | From the start to the end of recruitment at each participating site, approximately 4 weeks
  The number of staff volunteering to take part
Feasibility of study recruitment - the proportion of staff targeted through study advertising who volunteer to take part | From the start to the end of recruitment at each participating site, approximately 4 weeks
  The proportion of staff estimated to have been targeted through study advertising who volunteer to take part
Feasibility of study recruitment - the proportion of staff volunteering to take part in the study who are eligible | From the start to the end of recruitment at each participating site, approximately 4 weeks
  The proportion of staff volunteering to take part in the study who are eligible
Adherence to heart rate monitoring during 3-day lifestyle assessment | At Day 3 of the lifestyle assessment
  The proportion of time the heart rate monitor was worn by participants measured using data collected by the monitor
Adherence to completion of online journal during 3-day lifestyle assessment | At Day 3 of the lifestyle assessment
  The proportion of participants completing the journal
Feasibility of conducting interviews | On completion of interviews i.e. at approximately 8 weeks
  The proportion of participants in whom an interview is arranged and completed

SECONDARY OUTCOMES:
Heart rate variance | Measured during lifestyle assessment over a period of 3 days - at approximately 3 weeks post-recruitment
  Heart rate variance will be measured as a physiological indicator of stress via a heart rate monitoring device worn by each participant over a 3-day period.
Subjective mediators of stress | On completion of interviews i.e. at approximately 8 weeks
  Subjective mediators include personal, social and organisational factors identified through semi-structured interviews. Qualitative thematic analysis techniques will be used to identify individual and group characteristics and subjective mediators associated with periods of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Dippenaar, Principal Investigator — Anglia Ruskin University
Locations (1):
- Carmel Moore, Chelmsford, East of England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided